CLINICAL TRIAL: NCT03474497
Title: UCDCC#272: A Phase I/II Study of Intralesional IL-2, Hypofractionated Radiotherapy, and Pembrolizumab in Patients Refractory to Standard-of-Care PD-1/PD-L1 Checkpoint Blockade
Brief Title: UCDCC#272: IL-2, Radiotherapy, and Pembrolizumab in Patients Refractory to Checkpoint Blockade
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Megan Daly, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Megan Daly, MD, Associate Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1166212
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; Metastatic Melanoma; Metastatic Renal Cell Carcinoma; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Interleukin-2; pembrolizumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: All patients will receive pembrolizumab and intralesional IL-2 in combination with hypofractionated radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab/IL-2/Radiotherapy (Experimental): All patients will receive pembrolizumab and intralesional IL-2 in combination with hypofractionated radiotherapy.
  Interventions: Drug: IL-2; Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: IL-2 — • A total of four interleukin-2 treatments will be delivered into the treatment lesion by intralesional injection biweekly (at least 48 hours apart) starting 24-96 hours after the completion of radiotherapy and to be completed during the second on-trial cycle of Pembrolizumab. Intralesional injections will be performed by direct visualization and/or palpation of the lesion or under ultrasound or CT guidance as indicated.
Drug: Pembrolizumab — Pembrolizumab will be delivered at 200 mg in three week cycles per standard protocol.
Radiation: Radiotherapy — Radiotherapy will be delivered to the treatment lesion during the second cycle of therapy using an 8 Gy x 3 fractions palliative regimen. Fractions may be delivered on consecutive or every other day but must be completed during week 1-2 of cycle 2 and will not be repeated in future cycles.
  Other Names: Radiation Therapy

SUMMARY:
This is a phase I/II study that will evaluate the safety and toxicity of this combinatorial approach. Eligible patients >18 years of age with histologically proven metastatic NSCLC, melanoma, RCC, or HNSCC who have failed PD-1 / PD-L1 checkpoint blockade therapy will be enrolled. Patients must have a candidate treatment lesion (subcutaneous, nodal, or visceral) accessible and safe for radiotherapy and serial intralesional injections as specified by the protocol. They must also have at least one target lesion (distinct from treatment lesion and outside of treatment lesion radiation field) evaluable for response by RECIST.

This study will consist of a phase I dose escalation using a standard 3+3 design to determine safety and MTD of intralesional IL-2 which will be dose escalated in conjunction with standard fixed doses of RT and Pembrolizumab. At the MTD there will be a phase II dose expansion which will incorporate a simon-two stage design to assess efficacy and safety.

Patients will receive pembrolizumab and intralesional IL-2 in combination with hypofractionated radiotherapy.

DETAILED DESCRIPTION:
This is a phase I/II study that will evaluate the safety and toxicity of this combinatorial approach. Eligible patients >18 years of age with histologically proven metastatic NSCLC, melanoma, RCC, or HNSCC who have failed PD-1 / PD-L1 checkpoint blockade therapy will be enrolled. Patients must have a candidate treatment lesion (subcutaneous, nodal, or visceral) accessible and safe for radiotherapy and serial intralesional injections as specified by the protocol. They must also have at least one target lesion (distinct from treatment lesion and outside of treatment lesion radiation field) evaluable for response by RECIST.

This study will consist of a phase I dose escalation using a standard 3+3 design to determine safety and MTD of intralesional IL-2 which will be dose escalated in conjunction with standard fixed doses of RT and Pembrolizumab. At the MTD there will be a phase II dose expansion which will incorporate a simon-two stage design to assess efficacy and safety.

Patients will receive pembrolizumab and intralesional IL-2 in combination with hypofractionated radiotherapy.

* Radiotherapy will be delivered to the treatment lesion during the second cycle of therapy using an 8 Gy x 3 fractions palliative regimen. Fractions may be delivered on consecutive or every other day but must be completed during week 1-2 of cycle 2 and will not be repeated in future cycles.
* Pembrolizumab will be delivered at 200 mg in three week cycles per standard protocol.
* A total of four interleukin-2 treatments will be delivered into the treatment lesion by intralesional injection biweekly (at least 48 hours apart) starting 24-96 hours after the completion of radiotherapy and to be completed during the second on-trial cycle of Pembrolizumab. Intralesional injections will be performed by direct visualization and/or palpation of the lesion or under ultrasound or CT guidance as indicated.

Patients will be assessed by a physician once during the first week of radiotherapy, during each intralesional IL-2 injection, and with every cycle of pembrolizumab during the first three cycles. Thereafter patients will be assessed every 30 days during the study period and will continue until disease progression. All patients on active treatment will be discussed at weekly conferences of the trial investigators. Routine laboratory evaluation will occur pre-treatment and every 30 days. For response assessment patient will have imaging pre-treatment and after every three cycles of Pembrolizumab. For collateral studies patients will undergo mandatory treatment lesion biopsies and blood draws pre-treatment and during the needle placement for the final IL-2 treatment.

Preliminary efficacy as determined by abscopal response rate, ORR, DCR and PFS will be assessed every 3 cycles. The patient will remain on protocol treatment until progression as determined by irRECIST, treatment is no longer tolerated, or the patient has completed 12 months of treatment. Patients on active treatment at 12 months may continue to receive pembrolizumab but will revert to standard of care (SOC) management and be labeled in "follow up". At this time only PFS and long-term toxicity data will be collected every 3 months.

The primary endpoint is to determine if this regimen converts patients with resistance to PD 1/PD-L1 checkpoint blockade into responders as determined by abscopal response rate (defined as response rate at lesions not treated with RT + IL-2) using irRECIST as well as ORR, DCR, and PFS using RECIST 1.1. The secondary endpoint is tolerability, safety, and toxicity using CTCAE v4.03. Correlative studies include immunophenotyping serial tumor biopsies and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age with histologically proven metastatic NSCLC, melanoma, RCC, or head and neck SCC.
2. Failure to respond to checkpoint blockade therapy or previously responding patients who progress on PD-1/PD-L1 checkpoint blockade therapy.
3. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 - 1 (Appendix 1)
4. Presence of a candidate treatment lesion (subcutaneous or nodal lesions are preferable but visceral lesions will be considered) accessible and safe for radiotherapy and serial intralesional injections.
5. Presence of at least one target lesion (distinct from treatment lesion and outside of treatment lesion radiation field) evaluable for response by irRECIST
6. Life expectancy ≥ 6 months
7. Demonstrate adequate organ function as defined in Table 2, all screening labs should be performed within 10 days of treatment initiation.

   (Note: see protocol for table 2)
8. No other active malignancy.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Signed informed consent.
13. Ability to comply with the protocol.
14. Systolic ≥80.
15. No active auto-immune disease and not on therapy for auto-immune disease.
16. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible.

Exclusion Criteria:

1. Uncontrolled concomitant disease.
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Use of inhaled or topical steroids or systemic corticosteroids < 10 mg/ day is permitted.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) (excluding PD-1/PD-L1 inhibitor) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. History of severe autoimmune disease.
12. Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrollment (with the exception of checkpoint blockade therapy).
13. Treatment with systemic corticosteroids or other systemic immunosuppressive medications within past 4 weeks or 5 half-lives whichever is shorter. Use of inhaled or topical steroids or systemic corticosteroids < 10 mg/ day is permitted.
14. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
15. Has an active infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
21. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
22. Patients unable to tolerate checkpoint inhibitor therapy.
23. Unresolved Grade 3 or any grade 4 non-hematological, treatment-related AEs attributed to prior PD-1/ PD-L1 checkpoint blockade. A minimum of 2 weeks from prior PD-1/PD-L1 checkpoint blockade to initiating study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Daly, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UC Davis Medical Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-an-experimental-combination-of-injections-and-radiation-therapy-for-advanced-stage-solid-tumors-555849/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 3 (Starting Dose): Dose Level 3 (Starting dose):
  IL-2: Intratumoral, 3 x10^6 IU Tx 1, 7 x10^6 IU Tx 2, 15 x10^6 IU 7 x10^6 IU Tx 3-4 Radiation therapy: 8 Gy x 3 (week 1 of Cycle 2) Pembrolizumab: 200 mg q3 weeks (3w = 1 cycle)
- Dose Level 2: Dose Level 2:
  IL-2: Intratumoral, 3 x10^6 IU Tx 1, 7 x10^6 IU Tx 2-4 Radiation therapy: 8 Gy x 3 (week 1 of Cycle 2) Pembrolizumab 200 mg q3 weeks (3wk = 1 cycle)
- Dose Level 1: Dose Level 1:
  IL-2: Intratumoral, 3 x10^6 IU Tx 1-4 Radiation therapy: 8 Gy x 3 (week 1 of Cycle 2) Pembrolizumab 200 mg q3 weeks (3wk = 1 cycle)
- Dose Level -1: Dose Level -1:
  IL-2: Intratumoral, 1 x10^6 IU Tx 1-4 Radiation therapy: 8 Gy x 3 (week 1 of Cycle 2) Pembrolizumab 200 mg q3 weeks (3w = 1 cycle)
Period: Phase 1 dose finding
Arm/Group | Dose Level 3 (Starting Dose) | Dose Level 2 | Dose Level 1 | Dose Level -1
Started | 7 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Period: Phase 2 dose expansion
Arm/Group | Dose Level 3 (Starting Dose) | Dose Level 2 | Dose Level 1 | Dose Level -1
Started | 11 | 0 | 0 | 0
Completed | 11 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Abscopal Response Rate (ARR)
Description: To determine the abscopal response rate (ARR) defined as objective response rate (the number of patient that achieve a partial or complete response) at unirradiated sites using irRECIST criteria using imaging obtained every 60 days.
Time Frame: Up to time of response, about 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 14
Participants | 2

2. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) defined as the number of patients that achieve partial response (PR) or complete response (CR) per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions
Time Frame: Up to time of response, about 8.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 14
Participants | 2

3. Primary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) defined as the number of patients whose best overall response is either complete response (CR), partial response (PR) or stable disease (SD), as assessed by Response Evaluation Criteria in Solid Tumors Criteria version 1.1 (RECIST v1.1) for target lesions.
Time Frame: Up to about 10 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 14
Participants | 5

4. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) defined as the median time from initiation of study intervention to progressive disease, defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to about 7.3 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 15
months | 2.03 [1.8 to 7.3]

5. Secondary Outcome: Maximum Tolerated Dose (MTD) (Phase 1)
Description: To determine the maximum tolerated dose (MTD) of intralesional interleukin-2 (IL-2) that can be administered with hypofractionated radiotherapy (RT) and pembrolizumab.
Time Frame: Up to 90 days of treatment
Measure: Number; unit: x 10^6 International units (IU)
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 6
x 10^6 International units (IU) | 15

6. Secondary Outcome: Safety Profile and Toxicity
Description: Safety profile and toxicity of intralesional interleukin-2 (IL-2), radiotherapy (RT), and pembrolizumab defined as the number of patients experiencing treatment related adverse events (AE) grade ≥ 3, using CTCAE v4.03 (Common Toxicity Criteria for Adverse Events version 4.03,
Time Frame: Up to about 5.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
Number analyzed (Participants) | 18
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events assessed from first dose to 30 days after last treatment, approximately up to about 8 months. All-cause mortality assessed from first dose until death from any cause, approximately 5.5 years.
Arm/Group | Pembrolizumab/IL-2/Radiotherapy
All-Cause Mortality (participants affected / at risk) | 2/18
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab/IL-2/Radiotherapy (N=18)
Myocardial infarction (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Fever (General disorders) | 1
Rigors (General disorders) | 1
Sepsis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab/IL-2/Radiotherapy (N=18)
Anemia (Blood and lymphatic system disorders) | 2
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 4
General disorders and administration site conditions - Other, (General disorders) | 1
Infusion related reaction (General disorders) | 1
Injection site reaction (General disorders) | 4
Alkaline phosphatase increased (Investigations) | 2
Investigations - Other (Investigations) | 4
Lipase increased (Investigations) | 1
Lymphocyte count decreased (General disorders) | 6
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03474497/Prot_SAP_000.pdf